CLINICAL TRIAL: NCT06761599
Title: Frequency of Pulmonary Toxicity in Patients Treated for Hodgkin Lymphoma
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/046
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: group 1 — To determine treatment-induced pulmonary toxicity prevalence and risk factors in Hodgkin lymphoma patients during chemotherapy or radiation therapy.

SUMMARY:
Pulmonary toxicity during Hodgkin lymphoma treatment is significant for a variety of reasons, ranging from clinical care to therapeutic innovation and patient outcomes.

DETAILED DESCRIPTION:
Understanding chemotherapy-induced pulmonary issues, particularly bleomycin-induced toxicity, might enhance treatment efficacy, side effects, and quality of life for Hodgkin lymphoma patients. For Hodgkin lymphoma chemotherapy patients with pulmonary difficulties, which result in significant patient morbidity and mortality, early detection, proactive surveillance, and rapid management are required. Identifying the prevalence, risk factors, and clinical signs of pulmonary toxicity helps clinicians stratify treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Hodgkin lymphoma (HL) receiving treatment.
* Patients of all ages and both genders.
* Patients with histologically confirmed HL, as per the WHO 2016 classification.
* Patients who have undergone pulmonary function testing and assessment at specified time points during their treatment course.
* Patients with complete medical records documenting treatment regimens, including chemotherapy and radiotherapy details.

Exclusion Criteria:

* Patients with a diagnosis of another malignancy.
* Patients with incomplete medical records or missing data on treatment regimens and pulmonary function assessments.
* Patients with a history of significant pulmonary comorbidities, such as chronic obstructive pulmonary disease (COPD), interstitial lung disease, or pulmonary fibrosis, before HL diagnosis.
* Patients who are unable to complete pulmonary function tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: to check the Frequency of Pulmonary Toxicity in Patients Treated for Hodgkin Lymphoma
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
high-resolution computed tomography | 12 Months
  An HRCT (high-resolution computed tomography) scan is a type of CT scan healthcare providers use to get detailed images of your lungs. Providers most commonly use it to diagnose and monitor interstitial lung diseases and conditions that affect your small airways and alveoli (air sacs).

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Centre, 5-B, Sector A2, Phase 5, Hayatabad, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No